CLINICAL TRIAL: NCT06138392
Title: Clinical and Radiographic Performance of Early Loaded Dental Implants With a Conditioned Hydrophilic Surface: A Prospective Cohort Study With an 8.5- to 9.5-year Follow-up
Brief Title: Long-term Study in Early Loaded Hydrophilic Surface Implants
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Performance of early loading
Record Dates: First submitted 2023-10-10; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dental Implant
Keywords: Dental implant; Implant crowns; Hydrophilic implant surface; Early loading; Late implant placement
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental group
  Interventions: Device: Dental implant (ELEMENT RC INICELL, Thommen Medical)

INTERVENTIONS:
Device: Dental implant (ELEMENT RC INICELL, Thommen Medical) — Dental implant

SUMMARY:
Objective: To assess the clinical outcomes and patient satisfaction of early loaded implants with a hydrophilic, moderately rough surface for partially edentulous patients after a follow-up of 8.5 to 9.5 years.

Materials and methods: A prospective observational single-centre study involving 15 patients with single, delayed placement and early loaded implants in the posterior area was performed. Clinical and radiographical parameters, including biological and technical complications and patient satisfaction, were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18 and 75 years (inclusive)
* Partially edentulous patients with missing teeth in the posterior mandible (positions 34-37 and 44-47) and a healed site at least four weeks after tooth extraction
* Patients requiring a single dental implant
* Patients with physical status 1 or 2 according to the American Society of Anesthesiologists Classification System
* Inadequate native bone quality and quantity to place implants with a diameter of ≥4.0 mm
* Removable prosthesis or complete dentures in the antagonizing dentition
* Written informed consent

Exclusion Criteria:

* Patients with compromised general health contraindicating surgical intervention
* Presence of conditions requiring chronic routine prophylactic or prolonged use of antibiotics
* Heavy smokers (exceeding ten cigarettes/day or equivalent) and chewing tobacco users
* Pregnancy or childbearing potential with a positive urine pregnancy test
* Insufficient oral hygiene, untreated periodontitis (any residual pockets >4 mm), or persistent intra-oral infection
* Mucosal diseases such as erosive lichen planus
* Patients with severe bruxism or clenching habits
* Unwillingness to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated in an University Clinic
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance - survival | 10 years
  Survival was classified as the continued presence of both the implant and reconstruction in the mouth with no need of replacement and/or repair
Clinical performance - implant success | 10 years
  Implant success was classified as the absence of persisting subjective discomfort (patient compliance), lack of recurrent peri-implant infection with suppuration (European Federation of Periodontology 2018), absence of implant mobility on manual palpation, absence of any continuous peri-implant radiolucency at the radiological assessment.
Clinical performance - prosthetic success | 10 years
  Prosthetic success was defined as the absence of technical complications without needing any reconstruction repair.
Clinical performance - complications | 10 years
  A visual exploration of each implant and reconstruction was performed to detect any biological and technical complications.
Clinical performance - peri-implant health | 10 years
  During the clinical follow-up appointments, peri-implant health was evaluated by using a periodontal probe.
  Periodontal pockets (1-20) All parameters were evaluated mesially, distally, buccally, and orally in each implant; following the EFP guidelines (European Federation of Periodontology 2018).
Clinical performance - peri-implant health | 10 years
  During the clinical follow-up appointments, peri-implant health was evaluated by using a periodontal probe.
  Plaque index (1-3) All parameters were evaluated mesially, distally, buccally, and orally in each implant; following the EFP guidelines (European Federation of Periodontology 2018).
Clinical performance - peri-implant health | 10 years
  During the clinical follow-up appointments, peri-implant health was evaluated by using a periodontal probe.
  Bleeding on probing (yes/no) All parameters were evaluated mesially, distally, buccally, and orally in each implant; following the EFP guidelines (European Federation of Periodontology 2018).
Clinical performance - peri-implant health | 10 years
  During the clinical follow-up appointments, peri-implant health was evaluated by using a periodontal probe.
  Pus (yes/no) All parameters were evaluated mesially, distally, buccally, and orally in each implant; following the EFP guidelines (European Federation of Periodontology 2018).
Clinical performance - peri-implant health | 10 years
  During the clinical follow-up appointments, peri-implant health was evaluated by using a periodontal probe.
  Keratinized mucosa (mm) All parameters were evaluated mesially, distally, buccally, and orally in each implant; following the EFP guidelines (European Federation of Periodontology 2018).
Clinical performance - PIBL, implant-crown fit | 10 years
  To assess Peri-implant Bone Level (mm), a standardized digital periapical radiograph was taken at the scheduled follow-up visits.
  An independent examiner performed a radiological linear evaluation (mm) using image analysis software (ImageJ)
Clinical performance - PIBL, implant-crown fit | 10 years
  To assess implant-crown fit (misfit yes/no), a standardized digital periapical radiograph was taken at the scheduled follow-up visits.
  An independent examiner performed a radiological linear evaluation (mm) using image analysis software (ImageJ)
Clinical performance | 10 years
  Patient satisfaction with the implant treatment was evaluated using a 10 cm visual analogue scale (VAS). From 0 (The worst) to 10 (The best).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schimmel, Prof, Study Chair — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No